CLINICAL TRIAL: NCT03650543
Title: Effect of the CYP2C19 Polymorphism in Helicobacter Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Javeriana University (Other)
Collaborators: Universidad Nacional de Colombia (Other)
Responsible Party: Principal Investigator, Azucena Arévalo Galvis, MSc, Bacteriologist, Javeriana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00004554; 00004554 (Other Grant/Funding Number: Pontificia Universidad Javeriana); 12010U80401200 (Other: Pontificia Universidad Javeriana)
Record Dates: First submitted 2018-08-01; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: CYP2C19 Polymorphism; H.Pylori Infection; Therapy

STUDY DESIGN:
Intervention Model Description: A randomized single - blinded Clinical Trial conducted from 2012 to 2015 in Bogotá, Colombia. The aim was studying the effectiveness of triple therapy for H. pylori with amoxicillin, clarithromycin and standard dose of omeprazole versus amoxicillin, clarithromycin with dose of omeprazole according to CYP2C19 polymorphisms was studied, the subjects were allocated to a treatment regimen according to a randomized crossover sequence, provided by a computer-generated randomization list. Patients were contacted by telephone for assigned an appointment for treatment delivery according to the assigned group.
Who Masked: Care Provider
Masking Description: The mean masking was the treating Gastroenterologist doctor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- amoxicillin clarithromycin omeprazole 1 (Experimental): This group received triple standard therapy with standard doses of omeprazole. 20 mg "omeprazole" before breakfast and before dinner. 500 mg "clarithromycin" after breakfast and after dinner and 1 g "amoxicillin" after breakfast and after dinner for 10 days.
  Interventions: Drug: amoxicillin clarithromycin omeprazole 1
- amoxicillin clarithromycin omeprazole 2 (Experimental): This group received triple standard therapy, using 500 mg "clarithromycin" after breakfast and after dinner and 1 g "amoxicillin" after breakfast and after dinner for 10 days in addition with "omeprazole" but "omeprazole" doses were prescribed according to CYP2C19 genotype as a follows: a) Patients with CYP2C19 *1/*1 genotype (Early and ultrarapid Metabolizer): 40mg "omeprazole" before breakfast and before dinner. b) Patients with CYP2C19 *1/*2 or *1/*3 genotype (Intermediate Metabolizer): 20mg "omeprazole" before breakfast, 20mg before lunch and 20mg before dinner. c) Patients with CYP2C19 *2/*2 (Poor Metabolizer): 20mg "omeprazole" before breakfast and 20 mg before dinner.
  Interventions: Drug: amoxicillin clarithromycin omeprazole 2

INTERVENTIONS:
Drug: amoxicillin clarithromycin omeprazole 1 — Patients in this received triple standard therapy for eradication of H.pylori with standard doses of proton pump inhibitor (omeprazole), in combination with amoxicillin and clarithromycin in absence of antibiotic resistance.
  Other Names: Conventional therapy; Group 1
  Arms: amoxicillin clarithromycin omeprazole 1
Drug: amoxicillin clarithromycin omeprazole 2 — The treatment for patients in this group was prescribing triple standard therapy for H.pylori eradication with amoxicillin and clarithromycin in absence of antibiotic resistance but with different doses of proton pump inhibitor (omeprazole) according to CYP2C19 genotype in each patients.
  Other Names: Personalized therapy; Group 2
  Arms: amoxicillin clarithromycin omeprazole 2

SUMMARY:
Background: Triple therapy efficacy against Helicobacter pylori is low worldwide, thus alternatives must be sought to improve eradication. Aim: To determine CYP2C19 genetic polymorphism effect on H. pylori eradication.

Methods: A randomized single blinded clinical trial including 133 patients was carried-out. H. pylori infection was confirmed by histology and microbiological test. Antibiotic susceptibility to amoxicillin and clarithromycin was performed to avoid confusion bias in analysis results. CYP2C19 polymorphism "asterisk" *1, "asterisk"*2 and "asterisk" *3 was analyzed by Real time PCR (Roche ®), and nested PCR for CYP2C19 "asterisk" *17 polymorphism. Participants were randomized into two groups for different H. pylori therapies, one with standard omeprazole doses and another with omeprazole doses depending on CYP2C19 polymorphism. H. pylori eradicating was verified by stool antigen testing (Meridian ®). The general results was analysis by statistical computer program and the effectiveness of each therapy was analyzed by intention to treat (ITT) and by protocol (PP).

The study allowed to know the prevalence of the main polymorphisms of CYP2C19 in Bogotá-Colombia, also allowed to know the effectivenesses of the two therapies evaluated for H. pylori infection. Additionally, the importance of personalized medicine in H. pylori eradication therapy was known.

DETAILED DESCRIPTION:
Introduction:

H. pylori has been declared and ratified as carcinogen I by the World health organization (WHO) International agency for research on cancer (IARC). Globally first line therapy eradication treatment recommended for H. pylori, combines a proton-pump inhibitor (PPI) with two antibiotics (amoxicillin and clarithromycin or metronidazole). However, today effectiveness of this therapy is less than 75% "percentage", due mainly to H. pylori antibiotic resistance. Other factors involved in therapeutic failure are treatment adherence and host genetic factors that may affect medication pharmacokinetics, specifically PPI pharmacokinetics PPI play an essential role in eradication therapies, it suppresses deeply acid secretion, thus increasing hydrogen ion potential (pH) above 6.0. This allows H. pylori to replicate more actively than when stomach pH is less than 6.0, therefore improves antibiotic activity promoting greater antimicrobial agent stability and antibiotic concentration in stomach. PPIs action depends on its metabolism by cytochrome P450 (CYP) enzymes.Recent studies have showed that CYP2C19 genotype can affect PPIs ability to suppress acid secretion in the stomach, as has been observed for omeprazole. Omeprazole is metabolized by CYP2C19 (90%"percentage") and by CYP3A4 (10%"percentage"). CYP2C19 gene has 21 polymorphisms, three of which play an important role in PPIs metabolism. Thus, depending on polymorphism they are designated as early metabolizers (EM) ("asterisk"*1/"asterisk"*1), intermediate metabolizers (IM) ("asterisk"*1/"asterisk"*X) and poor metabolizers (PM) ("asterisk"*X/"asterisk"*X). Where "asterisk"*1 allele is the wild type allele ("Wild type") and "asterisk"*X correspond to mutated allele. Patients with genotype CYP2C19 "asterisk"*1/"asterisk"*2 o"asterisk" *1/"asterisk"*3 are IM and those with genotype CYP2C19 "asterisk"*2/"asterisk"*2 or CYP2C19 "asterisk"*3/"asterisk"*3 are PM. The presence of CYP2C19 "asterisk"*2 and CYP2C19 "asterisk"*3 polymorphisms predict the individual metabolizer phenotype. In 2006 the CYP2C19"asterisk"*17 allele was found, whose function is clinically important because heterozygotes, with CYP2C19"asterisk"*1/"asterisk"*17 forms are simply considered ultra-fast metabolizers by other authors. The clinical implication of this latter polymorphism relies on the following: if PPIs are quickly metabolized, standard PPIs dose fails to adequately suppress acid secretion, and H. pylori eradication therapy will be less effective if the microorganism is sensitive to antibiotics. A recent work in Colombia to eradicate H. pylori, using triple therapy with clarithromycin or levofloxacin combined with amoxicillin, reported that although the organism was sensitive to these antibiotics, there was variability with the achieved eradication. These results may suggest the possibility that additional factors, different from antimicrobial resistance, can influence the treatment effectiveness in our population.

General Methods:

The aim of present was to determine CYP2C19 genetic polymorphism influence on H.pylori eradication. For this purpose a randomized single blinded clinical trial was done. It was conducted from 2012 to 2015 in Bogotá, Colombia. The study was performed in accordance with Good Clinical Practice guidelines and ethical principles of the Declaration of Helsinki. Ethics Committee of the participating institutions approved the study protocol, where all participants signed written informed consent.

After obtaining informed consent, 356 patients were invited to participate in the study. All enrolled participants underwent initial endoscopy, carried-out at the upper endoscopy service, clinical center from Bogotá, D.C., Colombia to obtain gastric biopsy for histology, microbiological and genotypic test. However, due to the strict inclusion and exclusion criteria proposed, of the 356 participants, only 133 were included in the study.

All participants in the study underwent endoscopy of upper digestive tract under aseptic conditions, with a minimum of six hours of fasting. During the endoscopy five biopsies were taken from the antrum and four biopsies from the body for histopathology, microbiology and molecular analysis. For histopathological analysis, the biopsy samples were sent to pathology in separate properly marked containers. For microbiological and molecular analyses three antral and three body of the stomach biopsies were collected and used as follows: one biopsy from antrum for rapid urease test, two biopsies (antrum and one from the body of the stomach) for H. pylori culture and susceptibility test. Culturing was carried out only when one or both additional tests were positive for H. pylori. If the culture was negative, but any other tests were positive, microorganism detection was confirmed by molecular biology analysis (ureA gene detection H. pylori). It was considered a participant was infected with H. pylori when two or more tests were positive. Another biopsy was used for DNA extraction and subsequent analysis of CYP2C19 genetic polymorphism.

Culture was performed from biopsies of participants whose rapid urease test and histology were positive, from a biopsy of antrum and body of the stomach on Brucella agar (BD) enriched with 7% "percentage" v/v horse blood, Isovitalex (BD) and Helicobacter Pylori Selective Supplement (Dent) (Oxoid). Following, the samples were incubated at 37°C with 11% "percentage"carbon dioxide (CO2) for 3 to 5 days. Antibiotic susceptibility test from pure colonies was carried-out by agar dilution (gold standard method) according to the Clinical and Laboratory Standards Institute (CLSI) to determine amoxicillin and clarithromycin minimum inhibitory concentration (MIC). In addition, CYP2C19 polymorphism "asterisk"*1,"asterisk"*2,"asterisk"*3 and "asterisk"*17 were identified for all 133 patients included in this study. For this propose DNA was obtained from gastric biopsies by DNA Isolation from Human Samples from commercial Kit (QIAGEN), and then the identification of the respective polymorphisms was done.

CYP2C19 "asterisk"*1,"asterisk"*2,"asterisk"*3 polymorphisms were determined by real-time polymerase chain reaction (RT-PCR) using Modular Assays kit for human CYP2C19"asterisk"*2 and CYP2C19"asterisk"*3 (Roche), according to manufacturer's instructions. And nested PCR and Restriction Fragment Length Polymorphism (RFLP) was done for determination of allele "asterisk"*17 according with Baldwin et al. report.

Due to the study compared two types of therapies, the 133 patients were randomized for received the treatments into two groups by a computer program. Group one or conventional group and group 2 or personalized group. Both groups received amoxicillin and clarithromycin but first group received standard doses of omeprazole and in the second group omeprazole doses was adjusting according to the CYP2C19 polymorphism of each participant.

After performing microbiological and molecular testing, the participants were allocated to a treatment regimen according to a randomized crossover sequence, provided by a computer-generated randomization list. Participants were contacted by telephone for assigned an appointment for treatment delivery according to the assigned group.

All participants were given detailed information about the adverse effects that could occur with the different medications. Verification of possible adverse effects was performed telephonically using a validated and pre-coded questionnaire that included the following symptoms: diarrhea, metallic taste, nausea, bloated feeling, loss of appetite, vomiting, abdominal pain, constipation, and rash. The intensity of each symptom was graded from zero to three: 0: absent, 3: severe, using a Likert scale. Finally H. pylori eradication was verified 8 weeks post treatment by antigen test (Meridian®). For this test, each participants was requested a stool sample. The test was carried-out according to manufacturer's indications.

For the analysis of results, a database of the participants in excel and in spss was generated. These databases included general characteristics of each participant, result of each of the microbiology tests, molecular biology. Descriptive statistics and analysis of the effectiveness of the treatments used were carried out.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with functional dyspepsia or peptic ulcers
* Subjects between the ages of 19 and 70 years old
* Subjects who were referred for upper endoscopy, and had not received previous H. pylori eradication treatment within the last six months.
* Subjects who had not received anti-secreting acid, bismuth or antibiotics for other diseases 15 days before the endoscopy.
* For the study, only patients with sensitive isolates of H.pylori to amoxicillin and clarithromycin were included.

Exclusion Criteria:

* Patients with serious comorbidities.
* Pregnant women.
* Patients allergic to the medications used in this study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2012-09-10 (Actual); Primary Completion 2015-08-08 (Actual); Study Completion 2015-08-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness of each therapy by protocol (PP) | through study completion an average of 3 years
  Percentage

SECONDARY OUTCOMES:
Effectiveness of each therapy by intention to treat (ITT) | through study completion an average of 3 years
  Percentage

OTHER OUTCOMES:
Gender | through study completion an average of 3 years
  percentage of male and female
Weight | through study completion an average of 3 years
  Kilograms
Height | through study completion an average of 3 years
  centimeters
Body mass index | through study completion an average of 3 years
  kg/m^2
Prevalence of CYP2C19 polymorphism | through study completion an average of 3 years
  Percentage
Adverse effects in each therapy | through study completion an average of 3 years
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: Alba Alicia Trespalacios Rangel, Ph.D, Principal Investigator — Pontificia Universidad Javeriana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Sapone A, Vaira D, Trespidi S, Perna F, Gatta L, Tampieri A, Ricci C, Cantelli-Forti G, Miglioli M, Biagi GL, Paolini M. The clinical role of cytochrome p450 genotypes in Helicobacter pylori management. Am J Gastroenterol. 2003 May;98(5):1010-5. doi: 10.1111/j.1572-0241.2003.07427.x. PMID 12809821
- [Background] Sugimoto M, Furuta T, Shirai N, Kodaira C, Nishino M, Ikuma M, Ishizaki T, Hishida A. Evidence that the degree and duration of acid suppression are related to Helicobacter pylori eradication by triple therapy. Helicobacter. 2007 Aug;12(4):317-23. doi: 10.1111/j.1523-5378.2007.00508.x. PMID 17669104
- [Background] Furuta T, Graham DY. Pharmacologic aspects of eradication therapy for Helicobacter pylori Infection. Gastroenterol Clin North Am. 2010 Sep;39(3):465-80. doi: 10.1016/j.gtc.2010.08.007. PMID 20951912
- [Background] Scott D, Weeks D, Melchers K, Sachs G. The life and death of Helicobacter pylori. Gut. 1998 Jul;43 Suppl 1(Suppl 1):S56-60. doi: 10.1136/gut.43.2008.s56. PMID 9764042
- [Background] Furuta T, Shirai N, Sugimoto M, Nakamura A, Hishida A, Ishizaki T. Influence of CYP2C19 pharmacogenetic polymorphism on proton pump inhibitor-based therapies. Drug Metab Pharmacokinet. 2005 Jun;20(3):153-67. doi: 10.2133/dmpk.20.153. PMID 15988117
- [Background] Chaudhry AS, Kochhar R, Kohli KK. Genetic polymorphism of CYP2C19 & therapeutic response to proton pump inhibitors. Indian J Med Res. 2008 Jun;127(6):521-30. PMID 18765869
- [Background] Li-Wan-Po A, Girard T, Farndon P, Cooley C, Lithgow J. Pharmacogenetics of CYP2C19: functional and clinical implications of a new variant CYP2C19*17. Br J Clin Pharmacol. 2010 Mar;69(3):222-30. doi: 10.1111/j.1365-2125.2009.03578.x. PMID 20233192
- [Background] Furuta T, Sugimoto M, Shirai N, Ishizaki T. CYP2C19 pharmacogenomics associated with therapy of Helicobacter pylori infection and gastro-esophageal reflux diseases with a proton pump inhibitor. Pharmacogenomics. 2007 Sep;8(9):1199-210. doi: 10.2217/14622416.8.9.1199. PMID 17924835
- [Background] Isaza C, Henao J, Martinez JH, Sepulveda Arias JC, Beltran L. Phenotype-genotype analysis of CYP2C19 in Colombian mestizo individuals. BMC Clin Pharmacol. 2007 Jul 11;7:6. doi: 10.1186/1472-6904-7-6. PMID 17623107
- [Background] Arevalo-Galvis A, Trespalacios-Rangell AA, Otero W, Mercado-Reyes MM, Poutou-Pinales RA. Prevalence of cagA, vacA, babA2 and iceA genes in H. pylori strains isolated from Colombian patients with functional dyspepsia. Pol J Microbiol. 2012;61(1):33-40. PMID 22708344
- [Background] Baldwin RM, Ohlsson S, Pedersen RS, Mwinyi J, Ingelman-Sundberg M, Eliasson E, Bertilsson L. Increased omeprazole metabolism in carriers of the CYP2C19*17 allele; a pharmacokinetic study in healthy volunteers. Br J Clin Pharmacol. 2008 May;65(5):767-74. doi: 10.1111/j.1365-2125.2008.03104.x. Epub 2008 Feb 20. PMID 18294333
- [Background] Tang HL, Li Y, Hu YF, Xie HG, Zhai SD. Effects of CYP2C19 loss-of-function variants on the eradication of H. pylori infection in patients treated with proton pump inhibitor-based triple therapy regimens: a meta-analysis of randomized clinical trials. PLoS One. 2013 Apr 30;8(4):e62162. doi: 10.1371/journal.pone.0062162. Print 2013. PMID 23646118
- [Background] Sugimoto M, Furuta T. Efficacy of tailored Helicobacter pylori eradication therapy based on antibiotic susceptibility and CYP2C19 genotype. World J Gastroenterol. 2014 Jun 7;20(21):6400-11. doi: 10.3748/wjg.v20.i21.6400. PMID 24914361
- [Derived] Arevalo-Galvis A, Otero-Regino WA, Ovalle-Celis GN, Rodriguez-Gomez ER, Trespalacios-Rangel AA. Prevalence of CYP2C19 polymorphism in Bogota, Colombia: The first report of allele *17. PLoS One. 2021 Jan 27;16(1):e0245401. doi: 10.1371/journal.pone.0245401. eCollection 2021. PMID 33503046
- [Derived] Arevalo Galvis A, Trespalacios Rangel AA, Otero Regino W. Personalized therapy for Helicobacter pylori: CYP2C19 genotype effect on first-line triple therapy. Helicobacter. 2019 Jun;24(3):e12574. doi: 10.1111/hel.12574. Epub 2019 Mar 11. PMID 30859680